CLINICAL TRIAL: NCT07272889
Title: A Phase 1, Open-Label Study to Evaluate the Effect of Multiple Oral Doses of Bemnifosbuvir/Ruzasvir Fixed-dose Combination on the Single-Dose Pharmacokinetics of a Combined Oral Contraceptive (Ethinyl Estradiol/ Levonorgestrel) in Healthy Adult Female Participants of Non-Childbearing Potential
Brief Title: Drug-drug Interaction Study of Bemnifosbuvir/Ruzasvir (BEM/RZR) and Ethinyl Estradiol/Levonorgestrel (EE/LNG)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Atea Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AT-01B-012
Record Dates: First submitted 2025-11-19; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteer Study
MeSH Terms: interventions — Levonorgestrel; ruzasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- EE/LNG (Experimental)
  Interventions: Drug: Ethinyl Estradioll/Levonorgestrel (EE/LNG)
- BEM/RZR (Experimental)
  Interventions: Drug: Bemnifosbuvir/Ruzasvir (BEM/RZR)
- BEM/RZR + EE/LNG (Experimental)
  Interventions: Drug: Bemnifosbuvir/Ruzasvir (BEM/RZR) + Ethinyl Estradioll/Levonorgestrel (EE/LNG)

INTERVENTIONS:
Drug: Ethinyl Estradioll/Levonorgestrel (EE/LNG) — Treatment-A (EE/LNG): A single 0.03 mg/ 0.15 mg dose of EE/LNG (1 × 0.03 mg/ 0.15 mg tablet) will be administered in the morning under fasting conditions on Day 1.
  Other Names: Portia® 21
  Arms: EE/LNG
Drug: Bemnifosbuvir/Ruzasvir (BEM/RZR) — Treatment-B (BEM/RZR): A 550 mg/180 mg dose of BEM/RZR (2 × 275 mg/90 mg BEM/RZR FDC tablets) will be administered once daily (QD) under fasting conditions on Days 8 to 14.
  Other Names: BEM (AT-527)/RZR (AT-038)
  Arms: BEM/RZR
Drug: Bemnifosbuvir/Ruzasvir (BEM/RZR) + Ethinyl Estradioll/Levonorgestrel (EE/LNG) — Treatment-C (BEM/RZR + EE/LNG): BEM (550 mg)/ RZR (180 mg) as 2 × 275 mg/90 mg BEM/RZR FDC tablets will be administered QD in the morning under fasting conditions on Days 15 to 19. A single 0.03 mg/0.15 mg dose of EE/LNG (1 × 0.03 mg/ 0.15 mg tablet) will be concomitantly administered with BEM/RZR on the morning of Day 15.
  Other Names: BEM (AT-527)/RZR (AT-038); Portia® 21
  Arms: BEM/RZR + EE/LNG

SUMMARY:
Drug-drug interaction study between Ethinyl Estradioll/Levonorgestrel and Bemnifosbuvir/Ruzasvir

ELIGIBILITY:
Inclusion Criteria:

* Healthy post-menopausal or hormonally sterile female
* Minimum body weight of 50 kg and body mass index (BMI) of 18.0-30 kg/m2.
* Willing to comply with the study requirements and to provide written informed consent.

Exclusion Criteria:

* Infected with hepatitis B virus, hepatitis C virus, HIV or SARS-CoV-2.
* Abuse of alcohol or drugs.
* Use of other investigational drugs within 28 days of dosing.
* Concomitant use of prescription medications, or systemic over-the-counter medications.
* Other clinically significant medical conditions or laboratory abnormalities.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 24 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
PK of EE/LNG (Cmax) | Day 1,15
PK of EE/LNG (AUC) | Day 1,15

CONTACTS AND LOCATIONS:
Locations (1):
- Atea Study Site, Québec, Montreal, Canada